CLINICAL TRIAL: NCT00778596
Title: A Randomized, Double Blind Controlled Trial to Evaluate the Therapeutic Effect of Telbivudine With or Without Prednisolone Priming in Patients With Chronic Hepatitis B
Brief Title: Prednisolone Priming Study in Patients With Chronic Hepatitis B
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yun-Fan Liaw (Other)
Collaborators: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor-Investigator, Yun-Fan Liaw, Yun-Fan Liaw, Chang Gung Memorial Hospital
Organization: Chang Gung Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CST-L-1
Record Dates: First submitted 2008-10-21; First posted 2008-10-23 (Estimated); Last update posted 2012-05-25 (Estimated); Status verified 2012-05

CONDITIONS: Chronic Hepatitis B
Keywords: Hepatitis B; Telbivudine; Prednisolone
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — Prednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prednisolone priming (Experimental): Prednisolone priming 4 weeks, then treated with telbivudine.
  Interventions: Drug: Prednisolone
- Placebo priming (Placebo Comparator): Placebo priming for 4 weeks, then followed a telbivudine treatment for 2 years.
  Interventions: Drug: Placebo priming

INTERVENTIONS:
Drug: Prednisolone — Prednisolone priming for 4 weeks, then followed a telbivudine treatment for 2 years.
  Arms: Prednisolone priming
Drug: Placebo priming — Prednisolone priming for 4 weeks, then followed a telbivudine treatment for 2 years.
  Other Names: Placebo
  Arms: Placebo priming

SUMMARY:
Study purpose:

To investigate whether ALT rebound following corticosteroid priming enhances response to telbivudine therapy.

Efficacy assessments:

The primary endpoint will be the 1-year HBe-Ag seroconversion rate with or without prednisolone priming.

Data analysis:

A summary table will be presented as frequency tables for categorical variables as number, and percentage, whereas descriptive tables for continuous variables as number, mean ± SD and median (minimum, maximum). All statistical assessments will be two-sided and evaluated at significance level of 0.05. Continuous variables will be analyzed using t-test, or ANOVA, and categorical variables will be analyzed using chi-square or Fisher's exact test. A non-parametric method, Wilcoxon rank-sum or sign-rank tests will be conducted for continuous, and categorical variables if data is far from normal distribution.

DETAILED DESCRIPTION:
This is a Phase IV, multi-center, double-blinded, placebo control randomized study to evaluate the therapeutic effect of telbivudine with or without prednisolone priming in patients with chronic hepatitis B.

Patients are allocated to either group A or B randomly.

Group A: Patients initially receive a 4-week course of oral prednisolone (30 mg daily for 3 weeks and then 15 mg daily of 1 week). After a rest period of no treatment for 2 weeks, the patients receive telbivudine therapy at a daily dose of 600 mg for 2 years. Patients will be asked to come back to clinic for follow-up 6 months after telbivudine treatment.

Group B: Patients receive a 4-week course of placebo. After a rest period of no treatment for 2 weeks, the patients receive telbivudine therapy at a daily dose of 600 mg for 2 years. Patients will be asked to come back to clinic for follow-up 6 months after telbivudine treatment.

Eligible patients will be randomized prior to the first dose of study medication. The visit at which the patient receives the first dose will be defined as the study Baseline. Patients will return to the clinic at 3, 4, 6, 10, 14, 18, 30, 44, 58, 72, 86, 98, 110, 116, 122, 128 and 134 weeks post-Baseline. At each of these visits, routine clinical laboratory tests, adverse event inquiry, and other clinical assessments will be performed. Serum samples for HBV DNA analysis will be obtained at 4, 6, 30, 58, 86, 110 and 134 weeks. Serum samples for HBV sequencing will be obtained at Screening and Week 110 (or upon early termination from the study).

Complete physical examinations will be performed at each study visits to evaluate any adverse signs or symptoms reported by the patient.

Serum for HBeAg, antibody to HBeAg (HBeAb), HBsAg, and antibody to HBsAg (HBsAb) will be obtained at Screening, Baseline, and Weeks 6, 30, 58, 86, 110 and 134(or upon early termination from the study), and at all protocol-required follow-up visits.

Patients will be followed monthly for 6 months after discontinuation of study drug(s).

ELIGIBILITY:
Inclusion Criteria:

1. Treatment naïve patients or interferon-treated patients 6 months before, or oral antiviral agents treatment ≦ 2 weeks before or treatment < 3 months 1 year prior to screening.
2. Male or female, 18 to 65 years of age.
3. Documented chronic hepatitis B defined by all of the following:

   * Clinical history compatible with compensated chronic hepatitis B.
   * Detectable serum hepatitis B surface antigen (HBsAg) >6 months and at the screening visit.
   * Hepatitis B e antigen (HBeAg) positive >3 months.
   * Serum HBV DNA > 2x10^5 IU/mL and raised serum ALT > 2xULN but < 5xULN determined on at least 2 occasions 1 month apart before screen or within 3 months of pre-screen, raised serum ALT > 2xULN but < 5xULN determined 1 month apart before screen and at screen.4.
4. Liver biopsy showing chronic hepatitis and fibrosis stage ≦ 4 by Ishak classification within 6 months or fibrosis ≦ 4 between 6 to 12 months plus platelet count ≧ 150,000/mm3 or noninvasive assessment (fibroscan or ARFI) of liver fibrosis to excluding liver cirrhosis within 6 months.
5. Willing and able to comply with the study drug regimen and all other study requirements.
6. Willing and able to provide written informed consent to participate in the study.

Exclusion Criteria:

Patients will be excluded from the study for any of the following reasons:

1. Pregnant or nursing.
2. Of reproductive potential (men and women) and unwilling to use double-barrier method of contraception (i.e., condom with spermicide or diaphragm with spermicide).
3. Co-infection with hepatitis C virus (HCV), hepatitis D virus (HDV), or HIV.
4. History or clinical signs/symptoms of hepatic decompensation or portal hypertension, such as ascites, presence of esophageal varices or variceal bleeding, hepatic encephalopathy, or spontaneous bacterial peritonitis.
5. Liver cirrhosis (Ishak fibrosis score 5 or 6).
6. Any medical condition that requires prolonged or frequent use of systemic acyclovir or famciclovir (e.g., for recurrent herpes virus infections).
7. History of hepatocellular carcinoma (HCC) or findings suggestive of possible HCC, such as suspicious foci on imaging studies or elevated serum alpha-fetoprotein (AFP) levels. A history of treated malignancy other than HCC is allowable if the patient's malignancy has been in complete remission, off chemotherapy and without additional surgical intervention, during the preceding 3 years.
8. One or more known primary or secondary causes of liver disease other than hepatitis B (e.g., alcoholism, non-alcoholic steatohepatitis, autoimmune hepatitis, malignancy with hepatic involvement, hemochromatosis, alpha-1 antitrypsin deficiency, Wilson's disease, other congenital or metabolic conditions affecting the liver, congestive heart failure or other severe cardiopulmonary disease). Gilbert's syndrome and Dubin-Johnson syndrome will not exclude patients from participation in this trial.
9. History of clinically evident pancreatitis.
10. Currently abusing alcohol (i.e., an average daily intake of more than 40 g of ethanol) or illicit drugs or a history of alcohol abuse or illicit substance abuse within the preceding 2 years. Patients currently on methadone maintenance treatment programs are NOT eligible.
11. A medical condition that requires frequent or prolonged use of systemic corticosteroids (e.g., severe asthma, severe arthritis or autoimmune conditions, organ transplantation, adrenal insufficiency).
12. A medical condition requiring the chronic or prolonged use of potentially hepatotoxic drugs (dapsone, erythromycin, fluconazole, ketoconazole, rifampin, anti-tuberculosis regimens, etc.). All such drugs must have been discontinued ≥ 30 days prior to randomization.
13. A medical condition requiring use of nephrotoxic drugs (e.g., aminoglycosides, amphotericin B, foscarnet, vancomycin, cyclosporine, tacrolimus, or frequent nonsteroidal anti-inflammatory drugs (NSAIDS) or aspirin [administered daily for more than one week at a scheduled dose intended for anti-inflammatory therapy]). All such drugs must have been discontinued ≥ 30 days prior to randomization.
14. Any other concurrent medical or psychosocial condition likely to preclude compliance with the schedule of evaluations in the protocol or likely to confound the efficacy or safety observations of the study.
15. Enrolled or planning to enroll in another clinical trial of an investigational agent while participating in this study.
16. Any of the following laboratory values at Screening:

    * Hemoglobin (Hb) <11 mg/dL for men or <10 mg/dL for women.
    * Total white blood cell count (WBC) <2,500/mm3.
    * Absolute neutrophil count (ANC) <1,500/mm3.
    * Platelet count <75,000/mm3.
    * Serum albumin <3.2 g/dL.
    * Total bilirubin ≥2 mg/dL with direct bilirubin > 50% of total bilirubin.
    * Serum creatinine >1.0 x ULN.
    * Alpha-fetoprotein (AFP) >50 ng/mL (requires further evaluation, to rule-out hepatocellular carcinoma)
    * Creatinine clearance (CrCl) <0.83 mL/sec (<50 mL/min) calculated by the laboratory using the modified Cockcroft-Gault method.
    * Serum amylase or lipase ³1.5 x ULN.
    * Prothrombin time (PT) prolonged by >3 seconds or International Normalized Ratio (INR) > 1.5, based on the upper limits of normal (ULN) of the reference value, despite vitamin K administration.
17. Use of any investigational drugs within 30 days or 5 half-lives of randomization, whichever is longer.
18. Systemic malignancy within 5 years.
19. Previous treatment with telbivudine.
20. History of hypersensitivity to components of either telbivudine formulations, or to drugs with similar chemical structures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2009-02; Primary Completion 2012-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint will be the 1-year HBe-Ag seroconversion rate with or without prednisolone priming. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yun-Fan Liaw, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (4):
- Taiwan (4):
  - Chang Gung Memorial Hospital - Chiayi, Chiayi County
  - Chang Gung Memorial Hospital - Kaohsiung, Kaohsiung City
  - Chang Gung Memorial Hospital - Keelung, Keelung
  - Chang Gung Memorial Hospital, Linkou, Taoyuan County